CLINICAL TRIAL: NCT04412811
Title: A Prospective, Multicenter Survey of Cytomegalovirus (CMV) and Other Herpesviruses Infections and Diseases in Allogeneic Hematopoietic Stem Cell Transplant (allo-HSCT) Recipients.
Brief Title: Prospective Survey of CMV, Herpesviruses Infections and Diseases in Allo-HSCT
Acronym: CYTOALLOSURVEY
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Collaborators: Azienda Policlinico Umberto I (Other)
Responsible Party: Sponsor
Other Study IDs: CYTOALLO GITMO-AMCLI SURVEY
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hematologic Diseases; Stem Cell Transplant Complications; Cytomegalovirus Viremia; Herpesvirus Infection
Keywords: Haematopoietic transplantation, CMV, Herpesviruses
MeSH Terms: conditions — Hematologic Diseases; Herpesviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with hematological disease: Adult and children allogenic Hematopoietic stem cell transplantation recipients

SUMMARY:
Prospective observational study of epidemiological surveillance, multicenter, non-profit, spontaneous, Italian with objective to describe the incidence of CMV infections and diseases in adult and pediatric patients undergoing allo-HSCT during the first 6 months from transplant. This study will evaluate approximately 1500 subjects (with competitive enrolment) from GITMO investigational centers.

DETAILED DESCRIPTION:
This is a prospective observational study of epidemiological surveillance, multicenter, non-profit, spontaneous, italian on patients submitted to allogeneic haematopoietic stem cell transplantation organized under the auspices of the Gruppo Italiano Trapianti di Midollo Osseo that involves the principal Centres active in transplantation of any kind of hematopoietic stem cells in Italy.

Allogeneic haematopoietic stem cell transplantation patients continue to be one of the highest risk categories for developing viral infections. Cytomegalovirus infection is the leading viral cause of morbidity and mortality and HHV6 and EBV are other major causes of complications in transplant. The risk of these infections is directly related to the type of transplant.

A better and continuous monitoring of Cytomegalovirus and other herpesviruses complication in this setting would contribute to a better knowledge of the evolving epidemiology and would lead to a better use of diagnostic strategies and of preventive and therapeutic measures.

This study is aimed to identify epidemiological characteristics of allogeneic haematopoietic stem cell transplantation patients developing cytomegalovirus and other herpesviruses infections, risk factors, diagnostic peculiarities and factors that may guide to pre-emptive therapy versus prophylaxis strategies.

Virological monitoring and health care resources utilization in Allogeneic haematopoietic stem cell transplantation recipients according to the different risk of viral infection will be also assessed. This prospective analysis will provide useful information for local clinicians to define tailored antiviral strategies in line with the change of transplantation procedures.

All consecutive patients submitted to allogeneic haematopoietic stem cell transplantation will be prospectively monitored for Cytomegalovirus Cytomegalovirus, Herpesvirus human 6 and Virus Epstein-Barr infections and diseases during the six months from transplant, because most of viral infections and diseases occur within this period after transplant. Risk factors, incidence and prognostic factors of each viral infection and disease, as well as diagnostic and therapeutic strategies employed in the various transplant centers, will be evaluated in the overall population and in subpopulations according to different transplant characteristics.

The incidence of these infections and diseases will be also collected and described according to the different types of transplant and underlying disease conditions.

The Secondary Objectives are:

To assess the factors that may affect the incidence and the prognosis of allogeneic haematopoietic stem cell transplantation infections and diseases, as well as of Herpesvirus human 6 and Virus Epstein-Barr infections and related diseases To assess the impact of allogeneic haematopoietic stem cell transplantation infections and diseases on the overall and attributable mortality at 12 months from the transplant To describe the virological diagnostic strategies of allogeneic haematopoietic stem cell transplantation, Herpesvirus human 6 and Virus Epstein-Barr infections and the allogeneic haematopoietic stem cell transplantation specific immunological reconstitution tests used in the various centres To describe the antiviral strategies employed in the various centers and in the various subpopulations of transplant patients with focus on use of antiviral drugs in prophylaxis and therapy and use of allogeneic haematopoietic stem cell transplantation -specific intravenous IVIG in prophylaxis and therapy To evaluate the impact of a local strategy about use of antiviral drugs and allogeneic haematopoietic stem cell transplantation -specific IVIG in prophylaxis and therapy on the epidemiological findings, the clinical evolution of the allogeneic haematopoietic stem cell transplantation infections and diseases and on the Health Care Resources utilization (diagnostic procedures, pharmaco-utilization, hospitalization, outpatient visits).

A web system data entry will be used for this study. Data will be stored using specific e-CRFs designed by GITMO committee and includes mainly descriptive variables. Data Center will perform extensive consistency checks and issue electronic Query Forms in case of inconsistent data. Follow-up period for the evaluation of survival will be from the date of transplant until 12 months post-transplant or death. However, patients may not have 12 months follow up and if the patients are not having 12 months of observation due to lost to follow up and not due to mortality, these patients characteristics will be compared with the rest of the patients in order to ascertain there is no bias or estimate the bias.

The study will be conducted according to the principles of Good Clinical Practice, the current Italian and European laws and regulations, in agreement with the declaration of Helsinki. The protocol has been written and the study will be conducted according to The International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use Harmonized Tripartite Guideline for Good Clinical Practice, issued by the European Union. The responsible Local Ethical Committee approval must be obtained before starting the trial. A copy of the patient informed consent form must be submitted to the appropriate authority or committee, together with the protocol for written approval. Written approval of the protocol and informed consent by the responsible and appropriate authority or committee must be obtained prior to recruitment of patients to the study.

ELIGIBILITY:
Inclusion Criteria:

* Prospective observational study of epidemiological surveillance, multicenter, non-profit, spontaneous, Italian with objective to describe the incidence of CMV infections and diseases in adult and pediatric patients undergoing allo-HSCT during the first 6 months from transplant. This study will evaluate approximately 1500 subjects, with competitive enrolment from GITMO investigational centers.

Exclusion Criteria:

* Absence of consent Written information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and children allogenic Hematopoietic stem cell transplantation recipients
Sampling Method: Probability Sample
Enrollment: 1310 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Cytomegalovirus infection | 6 months from transplant
  incidence of Cytomegalovirus after allogeneic haematopoietic stem cell transplantation
Cytomegalovirus disease | 6 months from transplant
  incidence of Cytomegalovirus after allogeneic haematopoietic stem cell transplantation
Herpesvirus human 6 infection | 6 months from transplant
  incidence of human 6 infection after allogeneic haematopoietic stem cell transplantation
Herpesvirus human 6 disease | 6 months from transplant
  incidence of human 6 disease after allogeneic haematopoietic stem cell transplantation
Virus Epstein-Barr infection | 6 months from transplant
  incidence of Virus Epstein-Barr infections after allogeneic haematopoietic stem cell transplantation
Virus Epstein-Barr disease | 6 months from transplant
  incidence of Virus Epstein-Barr disease after allogeneic haematopoietic stem cell transplantation

SECONDARY OUTCOMES:
Overall Survival (OS) | These outcome measures will be assessed at 1 year from transplant
  OS is defined as the time from transplant to the date of death due to any cause or to the last date the patient was known to be alive (censored observation) or to the date of the data cut-off for final analysis
Disease Free Survival (DFS) | These outcome measures will be assessed at 1 year from transplant
  DFS is defined as the probability of being alive free of disease at any point in time.
Transplant Related Mortality (TRM) | These outcome measures will be assessed at 1 year from transplant
  TRM was defined as death due to any transplantation-related cause other than disease
Relapse risk (RR) | These outcome measures will be assessed at 1 year from transplant
  RR or risk ratio is the ratio of the probability of an outcome in an exposed group to the probability of an outcome in an unexposed group.
Acute Graft-versus-Host Disease | These outcome measures will be assessed at 100 days from transplant
  cumulative incidence of acute GvHD (grade II-IV)
chronic graft-versus-host disease | These outcome measures will be assessed at 1 year from transplant
  cumulative incidence and severity of chronic graft-versus-host disease

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Girmenia, Principal Investigator — Azienda Policlinico Umberto I
Locations (50):
- Italy (50):
  - Ospedale San Carlo, Potenza, Italy
  - Policlinico GB Rossi, Verona, Italy
  - UO Ematologia e TMO - Ospedale C. Panico, Tricase, Lecce
  - A.O.U. Policlinico Federico II, Napoli, Napoli
  - Fondazione IRCCS San Matteo, Pavia, Pavia
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - Ospedale Mazzoni, Ascoli Piceno
  - A.O.S. G. Moscati, Avellino
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - A.O.U. Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale San Orsola, Bologna
  - Ospedale Regionale Generale- Divisione Ematologia, Bolzano
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - Azienda Sanitaria Locale Br1 Ospedale "A. Perrino, Brindisi
  - CTMO PO "Businco" A.O. "G. Brotzu", Cagliari
  - Ospedale Ferrarotto, Catania
  - Struttura Complessa di Ematologia, Azienda Ospedaliera Santa Croce e Carle, Cuneo
  - Azienda Ospedaliera di Careggi, Florence
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, Foggia
  - AOU-IRCCS San Martino-IST, Genova
  - Ospedale Gaslini, Genova
  - Policlinico VIto Fazzi, Lecce
  - AOU Integrata, Mestre
  - Divisione di Ematologia - Istituto Nazionale dei Tumori, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Divisione Ematologia - Azienda Ospedaliera Universitaria - Policlinico -, Modena
  - Ospedale San Gerardo, Monza
  - AOU S. Giovanni di Dio e Ruggi D'Aragona, Napoli
  - Uoc Sit Tmo, Napoli
  - UOSC Ematologia con Trapianto CSE, AORN A. Cardarelli, AORN Cardarelli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - CTMO Osp. V. Cervello Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Azienda ospedaliera Universitaria di Parma, Parma
  - Policlinico San Matteo, Pavia
  - Ospedale S. Maria della Misericordia, Perugia
  - Dip. di Ematologia - Unità di Terapia Intensiva Ematologica per il Trapianto Emopoietico - Ospedale Civile di Pescara, Pescara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - Arciospedale S. M. Novella, Reggio Emilia
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Ospedale Bambin Gesù, Roma
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Roma
  - Dipartimento di Oncologia Medica ed Ematologia - Istituto Clinico Humanitas, Rozzano (MI)
  - Ospedale Moscati, Taranto
  - AOU CIttà della Salute e della Scienza, Torino
  - Ospedale Regina Margherita, Torino
  - A.O. Santa Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girmenia C, Chiusolo P, Marsili G, Piciocchi A, Mico MC, Greco R, Porto G, Galaverna F, Bonifazi F, Cutini I, Malagola M, Bramanti S, Busca A, Carella AM, Carotti A, Iori AP, Onida F, Bono R, Terruzzi E, Vacca A, Rinaldi A, Cavattoni IM, Picardi A, Faraci M, Lazzarotto T, Baldanti F, Clerici P, Castagna L, Martino M, Ciceri F. The Changing Impact of Human Cytomegalovirus Serology and Infection on Patient Outcome After Allogeneic Hematopoietic Stem Cell Transplantation: An Italian Prospective Multicenter Survey in the Era of Letermovir Prophylaxis. Open Forum Infect Dis. 2025 Apr 18;12(5):ofaf233. doi: 10.1093/ofid/ofaf233. eCollection 2025 May. PMID 40322267